CLINICAL TRIAL: NCT05643677
Title: Fruquintinib Plus Irinotecan Second-line Treatment for Advanced Gastric Cancer: a Single-arm, Open-label, Singer-center, Phase II Study
Brief Title: Fruquintinib Plus Irinotecan in the Treatment of Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xi Shi, archiater, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-E1-GC001
Record Dates: First submitted 2022-11-29; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib combined with irinotecan (Experimental): Fruquintinib combined with irinotecan as a second-line treatment for advanced gastric cancer
  Interventions: Drug: Fruquintinib; Drug: Irinotecan

INTERVENTIONS:
Drug: Fruquintinib — 4 mg PO, QD (3 weeks on, 1 week off)
  Other Names: Elunate
Drug: Irinotecan — participants will receive irinotecan, 100 mg/m2, intravenous drip, day1 and day 14 of every 4 weeks

SUMMARY:
This study explores the efficacy and safety of fruquintinib combined with irinotecan in the second-line treatment of patients with advanced gastric cancer, aiming to bring more second-line treatment options for patients with advanced gastric cancer.

DETAILED DESCRIPTION:
This study was a single-arm, open-label, single-center phase II study. A total of 47 patients with advanced gastric cancer who had previously failed standard first-line therapy were recruited to receive combined treatment with fruquintinib and irinotecan. The patients' progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR), overall survival (OS) and safety were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood this study and voluntarily signed informed consent;
2. ≥18 years old;
3. Histologically and/or cytologically confirmed metastatic or locally advanced gastric cancer or gastroesophageal conjunctive adenocarcinoma with at least one previous systemic therapy (note: Previous systemic treatment options approved by this protocol include single-drug or multi-drug combination chemotherapy or chemotherapy combined with immunotherapy, or failure of anti-HER-2 targeted therapy after positive HER-2);
4. At least one extragastric measurable lesion according to RECIST v1.1 criteria;
5. ECOG physical condition 0-1;
6. BMI≥18；
7. The expected survival time ≥12 weeks;
8. The functions of vital organs during the first 14 days of enrollment met the following requirements:

   * Neutrophil absolute count ≥1.5×109/L;
   * Platelet ≥80×109/L;
   * hemoglobin ≥90g/L;
   * Total bilirubin < 1.5 ULN;
   * ALT and AST < 2.5 ULN (< 5 ULN in patients with liver metastasis);
   * Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr)≥60ml/min;
   * endogenous creatinine clearance > 50ml/min;
9. Effective contraceptive measures should be taken by women of childbearing age or by men whose partners wish to have children;
10. Good compliance, cooperate with follow-up.

Exclusion Criteria:

1. Prior treatment with VEGF or VEGFR inhibitors;
2. Past treatment with irinotecan (However, patients who had previously received neoadjuvant or failed postoperative adjuvant therapy could be included as first-line therapy）;
3. Had participated in other drug clinical trials and received at least one drug therapy within 4 weeks prior to enrollment or had received other systemic antitumor therapy including chemotherapy, signal transduction inhibitors, immunotherapy, other investigational drugs;
4. Had other malignancies within 5 years prior to inclusion, except basal cell or squamous cell carcinoma of the skin after radical resection, or carcinoma in situ of the cervix;
5. The patient has a current disease or condition that affects drug absorption, or the patient is unable to take fuquinitinib orally;
6. Subjects who are allergic to the study drug or any of its adjuncts;
7. Electrolyte abnormalities identified by the investigator as clinically significant;
8. Hypertension that was not controlled by medication before enrollment was defined as: systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥100 mmHg;
9. Prior to enrollment, active gastric and duodenal ulcers, ulcerative colitis and other digestive diseases, active bleeding in unresectable tumors, or other conditions that researchers determined may cause gastrointestinal bleeding and perforation;
10. Patients with significant evidence or history of bleeding tendency within 3 months prior to enrollment (bleeding within 3 months>30 mL, hematemesis, black feces, hematochezia), hemoptysis (within 4 weeks>5 mL fresh blood) or a thromboembolic event (including stroke and/or transient ischemic attack) within 12 months;
11. History of severe cardiovascular and cerebrovascular diseases:

    * Cerebrovascular accident (excluding lacunar infarction, mild cerebral ischemia or transient ischemic attack), myocardial infarction, unstable angina, and poorly controlled arrhythmia (including QTc interval ≥450ms for male and 470 ms for female) within 6 months before the first administration of the study drug (QTc interval ≥ 490ms for female) Fridericia formula);
    * New York Heart Association (NYHA) Cardiac Function Rating > Grade II or left ventricular ejection fraction (LVEF) < 50%;
12. Clinically uncontrolled active infections, such as acute pneumonia, active hepatitis B or C (previous history hepatitis B virus infection regardless of drug control, hepatitis B virus DNA≥1×104 copies /mL or > 2000 IU/ml);
13. Symptomatic brain or meningeal metastases (except those with brain metastases that have undergone local radiotherapy or surgery for more than 6 months and whose disease control is stable);
14. Women who are pregnant (tested positive for pregnancy before medication) or who are breastfeeding;
15. Two consecutive urine routine tests indicated urine protein ≥2+, and the 24-hour urine protein volume was reexamined > 1.0g;
16. Patients with clinical symptoms of ascites or pleural effusion;
17. The patients were not considered suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS was defined as the time from randomization until the date of first occurrence of investigator-assessed radiological disease progression or death due to any cause, whichever came first.

SECONDARY OUTCOMES:
Objective remission rate (ORR) | up to 12 months
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and kept for a certain time, including cases of complete remission and partial remission.
Disease control rate (DCR) | up to 12 months
  The percentage of patients whose tumors shrink or stabilize for a certain amount of time. DCR is the sum of complete, partial response and stable rate, that is, DCR=CR+PR+SD.
Overall survival（OS） | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  OS was defined as the time from the date of randomization to the date of death due to any cause. For subjects who were alive or lost to follow-up by the data analysis cut-off date, survival was censored at the subject's last known survival time.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Shi, Principal Investigator — First Affiliated Hospital of Fujian Medical University